CLINICAL TRIAL: NCT06635174
Title: Efficacy of 50% Oral Dextrose As Pain Relief in Newborns Before Bladder Catheterization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Ali Redha Taqi Al Qubtan, emergency resident, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OmanMedAQ
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pain Management; Neonatal Pain
Keywords: 50% dextrose; neonatal pain management
MeSH Terms: conditions — Agnosia | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Total of 90 patient divided randomly in 2 groups, one group will receive 2ml of 50% oral dextrose and control group will receive 2ml of normal water as placebo. The Neonatal Infant Pain Scale (NIPS) will be used to measure the pain score among the infants. It was designed and validated in Canada by Lawrence J Alcock D et al. It uses the behaviors that nurses have described as being indicative of infant pain or distress. It is composed of six (6) Parameters Facial expression Cry Breathing patterns Arms Legs State of arousal
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be generated at the local pharmacy by a computer program in blocks of two and the randomization allotment only will be known by a pharmacist not involved in the care of the children.
  after that the pharmacist will prepper the syringe than contain the 2ml 50% dextrose or the placebo 2ml normal water. each syringe will have code. the code key will be only with the pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): in this arm participant will receive oral 2ml of normal water
  Interventions: Other: normal water
- 50% dextrose group (Experimental): this arm will include the participant who will receive 50% oral dextrose
  Interventions: Other: Dextrose

INTERVENTIONS:
Other: Dextrose — we are using 2ml of 50% dextrose
  Arms: 50% dextrose group
Other: normal water — patient will receive 2ml of normal water
  Arms: control group

SUMMARY:
The aim of this study is to determine the effect of 50% oral dextrose in reducing pain before Bladder Catheterization.

This study will answer the following question

Is there any effect of 50% dextrose in reducing pain response to infants from age 1-90 days undergoing bladder catheterization during their visit in emergency department it is double blind randomized control trial comparing 2ml 50% dextrose as oral solution with placebo 2ml of normal water

Primary Objective

- To evaluate the impact of administrating oral glucose on pain control compared with placebo in blood pressure , Heart rate, respiratory rate and oxygen saturation before and after the procedure

Secondary Objectives

* To compare random blood sugar before and after the procedure
* To compare the incident and the duration of crying in both groups

administration of oral solution 2ml of solutions to be administered orally as drops at tip of the tongue after that will wait for 2 minutes before the procedure start , after 2 minutes from the oral solution , the procedure will start

DETAILED DESCRIPTION:
During first days of the life of New-borns, they go through a lot of painful procedures such as blood tests and immunizations that lead to painful experiences and distress. For long period of time it was believed that young children do not feel the painful stimuli. Recent studies have proven that they have all the anatomical, physiological and neurochemical system to feel for the pain (1). In fact, they have low threshold for the pain stimuli due to immature suppressive mechanism (2). There are several consequences that pain can cause to children such as: respiratory distress, changes in the metabolic and intracranial system, induce significant behavioural reactions and increase sensitivity to pain.

For these reasons, as well as for ethical reasons, it is advisable to find an acceptable method to reduce pain and distress during painful procedures. Pharmacologic treatment is not recommended for New-borns with acute, recurring, and short-term painful procedures. Studies has reported an alternative way which can be used for pain relive such as using oral sweeteners (3). World-widely, national and international guidelines recommended the use of oral sweeteners such as Sucrose and glucose before painful procedures (4). Researchers found that administration of oral dextrose can raise the pain threshold by activating endogenous opioids (5). The maximum effect can be observed at 2 minutes after administration (6). It is not clear what is the exact effective dose that can be used during painful procedure (7). Several studies used 2ml of dextrose, but other studies have reported an effect with 0.05 mL (8).

Study done by thyr et al (9) shows sweet solution can be used as a simple and safe method to reduce the distress following immunization in infants up to 12 months. A systematic review by Harrison et al (10) reported that Infants aged 1-12 months received oral sucrose or glucose before immunization had moderately reduced incidence and duration of crying.

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 day to 90 days
* Did not received analgesia for last 6 hours

Exclusion Criteria:

* Preterm newborns presenting in ED younger than 38 weeks (corrected age)
* Unstable child
* Suspicion of enterocolitis
* Esophageal- tracheal fistula not operated
* Known case of fructose intolerance
* Oral congenital malformation (cleft palate)

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
change in blood pressure | 3 minutes, 5 minutes and 7 minutes after oral solution will be administrated
  blood pressure will be measured before the procedure and 3 minutes, 5 minutes and 7 minutes after oral solution administration. each vital will be analyzed as single variable comparing it with the baseline.
  for example (baseline blood pressure will be compared with the blood pressure during procedure after oral solution) the different of both blood pressure will be analyzed whiter there is significant change or not in both group
change in The Neonatal Infant Pain Scale (NIPS) | 3 minutes, 5 minutes and 7 minutes after administration of oral solution
  the Neonatal Infant Pain Scale (NIPS) will be calculated by trained treating nurse staff 3 minutes, 5 minutes and 7 minutes after administration of oral solution
change in the heart rate | 3 minutes, 5 minutes and 7 minutes after oral solution administration.
  heart rate will be measured before the procedure and 3 minutes, 5 minutes and 7 minutes after oral solution administration. each vital will be analyzed as single variable comparing it with the baseline.
  for example (baseline heart rate will be compared with the heart rate during procedure after oral solution) the different of both heart rate will be analyzed whiter there is significant change or not in both group
change in respiratory rate | 3 minutes, 5 minutes and 7 minutes after oral solution administration.
  respiratory rate will be measured before the procedure and 3 minutes, 5 minutes and 7 minutes after oral solution administration. each vital will be analyzed as single variable comparing it with the baseline.
  for example (baseline respiratory rate will be compared with the respiratory rate during procedure after oral solution) the different of both heart rate will be analyzed whiter there is significant change or not in both group

SECONDARY OUTCOMES:
random blood sugar | 10 minutes
  the random blood sugar of the patient will be compared before and after administration of oral solution
the duration of crying in placebo group | 10 minutes
  the duration of crying in placebo group will be calculated from time of starting procedure to the time in which child will stop crying
the duration of crying in dextrose group | 10 minutes
  the duration of crying in dextrose group will be calculated from time of starting procedure to the time in which child will stop crying

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Al Qubtan, Muscat, Muḩāfaz̧at Masqaţ, Oman

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in randomized control trials. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- See also: Related Info — https://pubmed.gov